CLINICAL TRIAL: NCT04925349
Title: MATRIX - "Modeling Macrophages Activation Pattern in X-linked Adrenoleukodystrophy, Metachromatic Leukodystrophy and Adult Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia"
Brief Title: Modeling Macrophages Activation Pattern in X-linked Adrenoleukodystrophy, Metachromatic Leukodystrophy and Adult Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia
Acronym: MATRIX
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190197; IDRCB (Other: 2019-A00087-50)
Record Dates: First submitted 2019-04-15; First posted 2021-06-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Adrenoleukodystrophy; Adrenomyeloneuropathy; Metachromatic Leukodystrophy; Adult-Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia
Keywords: Leukodystrophy; Central Nervous System Diseases; Nervous System Diseases; Immune system; Neuroinflammation
MeSH Terms: conditions — Adrenoleukodystrophy; Leukodystrophy, Metachromatic; Hereditary Diffuse Leukoencephalopathy with Spheroids; Central Nervous System Diseases; Nervous System Diseases; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample for MAC analyses and blood sample for blood cells count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- affected subjects: * adult patients with adrenomyeloneuropathy/adrenoleukodystrophy
  * children with adrenoleukodystrophy
  * children with metachromatic leukodystrophy
  Interventions: Diagnostic Test: Blood sample collection
- control subjects: * healthy children
  * heatthy adults
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — blood sample collection

SUMMARY:
This study is a national, non-randomized, open-label, multi-site with minimal risk study in adult with adrenomyeloneuropathy (AMN), childhood and adult subjects with cerebral ALD (cALD), juvenile/adult metachromatic leukodystrophy (MLD) and adults with leukoencephalopathy and axonal spheroids and pigmented glia (ALSP). 49 subjects will be enrolled with one blood sample collection during one of their medical follow-up visit.

This trial will evaluate the role of innate immunity to influence disease progression in X-ALD, MLD and ALSP, and if the mutations related to these leukodystrophies result in a specific immune response leading to the pathogenesis.

DETAILED DESCRIPTION:
X-linked Adrenoleukodystrophy (X-ALD), Metachromatic Leukodystrophy (MLD) and Adult-onset leukoencephalopathy with axonal spheroids and pigmented glia (ALSP) are among the most frequent inherited leukodystrophies. X-ALD and MLD can affect both children and adults, while it is thought that ALSP onset exclusively during adulthood. These three diseases are characterized by phenotypic variability and poor genotype-phenotype correlation. In childhood forms of MLD and childhood cerebral ALD (C-CALD) a devastating cerebral demyelination and neuronal degeneration lead to a rapid neurologic degradation and premature death. Patients with the adult form of X-ALD (adrenomyeloneuropathy (AMN), 60% of males) display a progressive spastic paraplegia without brain involvement. However, 20% of AMN patients will also develop cerebral ALD. Patients diagnosed with the juvenile/adult (JA-) MLD form are affected by a progressive decline of their cognitive function, followed later by that of the motor abilities. ALSP patients present a rapidly progressive neurodegenerative disorder that impairs behavioural, cognitive and motor functions.

Several arguments support the contribution of the immune response and neuroinflammation in these three leukodystrophies. In X-ALD, activation of microglia (macrophages of the CNS) plays an essential role in the acute demyelination phase, where a severe inflammatory process occurs. In ALSP, the dysfunctional protein (CSF1R) is almost exclusively expressed in microglia. Even if MLD is not considered as a neuroinflammatory disease per se, microglia activation and increased inflammatory cytokines are observed in the brain of MLD patients and mice. Even if the most commonly accepted hypothesis is that neuroinflammation is caused by secondary activation of microglia following phagocytosis of myelin debris full of undegraded material, a primitive role of the inflammation due to macrophages (MAC) dysfunction has emerged in recent years.

MATRIX proposes to explore how disease-related mutations affect key components of MAC activation responses and how it reflects on their functionality.

ELIGIBILITY:
Inclusion Criteria:

Boys aged between 3 and 18 years (inclusive) diagnosed with C-CALD (elevated levels of VLCFA and leukodystrophy at brain MRI)

* Boys or girls aged between 15 months and 18 years (inclusive) diagnosed with MLD (low ARSA activity and accumulation of sulfatides in urine)
* Presymptomatic boys carrying ABCD1 mutations aged between 3 and 18 years (inclusive) (PRE-ALD)
* Adult males or females aged between 18 and 60 diagnosed with MLD (low ARSA activity and accumulation of sulfatides in urine)
* Males aged between 18 and 60 years diagnosed with AMN (elevated VLCFA and clinical symptoms of AMN without leukodystrophy at brain MRI)
* Males aged between 18 and 60 years diagnosed with CALD (elevated VLCFA with leukodystrophy at brain MRI)
* Adult males or females aged between 18 and 60 years diagnosed with ALSP (CSF1R mutation and leukodystrophy at brain MRI)
* Presymptomatic patient adults (males or females) carrying CSF1R mutations (PRE-ALSP)
* Children (15 months-18 years) without neurologic disease (no obvious neurological symptoms, normal neurologic examination)
* Adults aged between 18 and 60 years without neurologic disease (no overt neurological symptoms)
* Informed consent obtained :
* from the parents or guardian for children patients and children controls;
* from subject himself for adult patients and adult controls.

Exclusion Criteria:

* Participation to a therapeutic clinical trial
* Treatment likely to modify the immune system
* Unable to have a blood collection (i.e. low hemoglobin level at the investigator's judgment)
* Any other reason, to the discretion of the investigator
* Children or adults without health insurance or social security

Ages: 15 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric and adult populations. Both affected (C-CALD, AMN, A-CALD, MLD, ALSP), presymptomatic children carrying ABCD1 mutations (PRE-ALD), presymptomatic patient adults carrying CSF1R mutations (PRE-ALSP) and age-matched control subjects will be enrolled (N=10/group). Minor subjects (C-CALD, MLD, PRE-ALD and controls) will be included, based on childhood onset of C-CALD and MLD
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Macrophages functionality - distribution of monocytes | 2 years after blood collection
  distribution of monocytes in the CD14-/+/++ and CD16-/+ classification using flow cytometry (% of CD14++/16-; CD14++/16+; CD14+/16+; CD14-/16-)
Macrophages functionality - myelin phagocytosis capacity | 2 years after blood collection
  percentage of myelin high, myelin low and myelin negative cells using flow cytometry
Macrophages functionality - HLA levels | 2 years after blood collection
  maximum fluorescence intensity for HLA markers using flow cytometry

SECONDARY OUTCOMES:
Macrophages metabolic profiling | 2 years after blood collection
  Macrophages metabolic profiling (>2000 metabolites) using liquid chromatography coupled to high resolution mass spectrometry
Macrophages transcriptomic profiling | 2 years after blood collection
  Macrophages transcriptomic profiling (>1200 coding and non coding genes) : RNA sequencing using NextSeq 500 Illumina (60 million single-end, 150 base reads ) and analysis (using FastQC, Picard-Tools, Samtools and rseqc softwares

CONTACTS AND LOCATIONS:
Overall Officials: Fanny MOCHEL, MCU-PH, Principal Investigator — Institut du Cerveau et de la Moëlle épinière; Violetta ZUJOVIC, PhD, CR1, Study Chair — Institut du Cerveau et de la Moëlle épinière; Caroline SEVIN, PhD, Study Director — Kremlin Bicêtre Hôpital
Locations (2):
- France (2):
  - AP-HP Hôpital Bicêtre, Le Kremlin-Bicêtre
  - AP-HP Hôpital La Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miron VE, Boyd A, Zhao JW, Yuen TJ, Ruckh JM, Shadrach JL, van Wijngaarden P, Wagers AJ, Williams A, Franklin RJM, Ffrench-Constant C. M2 microglia and macrophages drive oligodendrocyte differentiation during CNS remyelination. Nat Neurosci. 2013 Sep;16(9):1211-1218. doi: 10.1038/nn.3469. Epub 2013 Jul 21. PMID 23872599
- [Background] Weinhofer I, Zierfuss B, Hametner S, Wagner M, Popitsch N, Machacek C, Bartolini B, Zlabinger G, Ohradanova-Repic A, Stockinger H, Kohler W, Hoftberger R, Regelsberger G, Forss-Petter S, Lassmann H, Berger J. Impaired plasticity of macrophages in X-linked adrenoleukodystrophy. Brain. 2018 Aug 1;141(8):2329-2342. doi: 10.1093/brain/awy127. PMID 29860501
- [Background] Berger J, Forss-Petter S, Eichler FS. Pathophysiology of X-linked adrenoleukodystrophy. Biochimie. 2014 Mar;98(100):135-42. doi: 10.1016/j.biochi.2013.11.023. Epub 2013 Dec 4. PMID 24316281
- [Background] Gieselmann V, Krageloh-Mann I. Metachromatic leukodystrophy--an update. Neuropediatrics. 2010 Feb;41(1):1-6. doi: 10.1055/s-0030-1253412. Epub 2010 Jun 22. PMID 20571983